CLINICAL TRIAL: NCT06781021
Title: The Effect of Tranexamic Acid Vs Torniquet on Visual Clarity in Knee Arthroscopic Anterior Cruciate Ligament (ACL) Reconstruction
Brief Title: The Effect of Tranexamic Acid Vs Torniquet on Visual Clarity in Knee Arthroscopic ACL Reconstruction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREC-MN.049,2023/2024
Record Dates: First submitted 2024-11-19; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: ACL Tears
Keywords: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Tourniquets

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: All patients will be positioned supine and administered spinal anesthesia. In all cases the application of a pneumatic torniquet will be applied to the proximal thigh after induction of anesthesia but will not be inflated for the group receiving TXA. Dependent on the randomized groups assigned; The standard torniquet pressure of 300 mm Hg will only be inflated for persons assigned to the torniquet group who will receive normal saline intravenously. Only the research assistant and the anesthetic staff will be aware of whether inflation of torniquet was applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tourniquet Surgery (Active Comparator): Torniquet surgery prevents blood loss by acting as a physical barrier to cut vessels and tissue. This physical barrier is in the form of pressure which is applied to the vessels but also to the surrounding tissues it touches. This pressure can damage nerves, muscle which can delay return to normal function afterwards if applied for a prolonged period. This however has not been a common occurrence and is used as the standard of care in ACL arthroscopic surgeries.
  Interventions: Procedure: Tourniquet; Procedure: TXA
- TXA Surgery (Active Comparator): TXA does the has the same function without the physical compression. In other words, it acts as a chemical torniquet. It enables clotting at damaged tissue which are more likely to bleed and obstruct the surgical field. This drug has not been shown to have any adverse reactions and is safe for use.
  Interventions: Procedure: Tourniquet; Procedure: TXA

INTERVENTIONS:
Procedure: Tourniquet — In all cases the application of a pneumatic torniquet will be applied to the proximal thigh after induction of anesthesia but will not be inflated for the group receiving TXA.
Procedure: TXA — In all cases the application of a pneumatic torniquet will be applied to the proximal thigh after induction of anesthesia but will not be inflated for the group receiving TXA.

SUMMARY:
Study Objective: The study aims to determine if tranexamic acid (TXA) is as effective as a tourniquet in improving visual clarity during arthroscopic ACL reconstruction surgery.

Study Design: This is a randomized prospective controlled trial involving patients with complete ACL tears. Participants will be randomly assigned to either receive TXA or undergo surgery with a tourniquet.

Data Collection: The study will use questionnaires and scales to assess the effects of TXA on visual clarity. Data will be stored securely and analyzed using the SPSS system.

Ethical Considerations: Ethical guidelines will be strictly followed, including informed consent, confidentiality, and the right to withdraw from the study at any time without affecting the standard of care.

Expected Outcome: The study aims to provide insights into the efficacy of TXA in improving surgical visibility, potentially influencing future protocols in arthroscopic surgeries. Results will be disseminated through academic presentations and publications.

DETAILED DESCRIPTION:
Study Design This study is a randomized prospective controlled trial. All patients with complete ACL from the three orthopedic teams at UHWI will be screened for inclusion criteria ACL tears requiring reconstruction for the first time. Patients will be approached by the Research Assistant and once agreement to participate has been obtained, will be informed of the study and given an informed consent (Appendix A). All consents will be done by the Research Assistant not involved in patient care.

The recruitment will take place in a discrete room within Orthopedics outpatient department where the patient will be informed of the details of the study and the right to participate or refuse. It will be reinforced that refusal to participate will not void the standard of care offered to patient. The study will be conducted over a two (2) year period in the Main Operating Theatre. The information gathered will be stored on a password encrypted computer stored in the Principal Investigator's office which can be accessed only by the Investigator or Principal Investigator. Data will be analyzed using Statistical Package for the Social Sciences (SPSS)

Meta analysis and subsequent prospective randomized studies have estimated that tourniquet use would be expected to be associated with poor visibility in only 0-3% of arthroscopic knee procedures. Excellent visibility would be expected in 90% to 97% of cases while no tourniquet would produce good or excellent visibility in approximately 80% of procedures (36, 37). A construct of 2 pairs of simulation populations with a) 97% scores of 1 (excellent visibility) in both the control and experimental groups and b) 97% scores of 1 in the control group and 80% scores of 1 in the experimental group. When the two populations with no stochastic difference were sampled, a sample size of 30 per arm was adequate to produce a BF_10 greater than 3 (i.e. support for the alternate hypothesis) for 90% of samples. Conversely, for two populations where there is a stochastic superiority of the control to the experimental, a sample size of 20 per arm produces a BF_10 less than 1/3 (i.e. support for the null hypothesis) for 90% of samples. We will be analyzing on an incremental basis and stop patient accrual when we either achieve a BF_10 greater than 10 or less than 1/10 (strong evidence for the alternate or null hypothesis) (35) or we achieve a cumulative sample size of 60 patients.

Research Procedures/Protocols - Data Collection/Research Intervention Procedures

Patients will be randomized with the help of an online randomization tool Randomization tool @ https://ctrandomization.cancer.gov/tool/ (National Cancer Institute Clinical trial randomization tool) being placed in one of two arms: TXA alone and Torniquet alone.

Patient Recruitment A flyer (Appendix A) will be placed at strategic areas (e.g. cashiers, radiology department, physiotherapy department) advertising the study. Patients will be seen in the Outpatient orthopedic clinic and once the diagnosis of a Complete ACL tear is made, the patients will be recruited by the Research Assistant who is aware of the protocols and nature of study. The recruitment will continue until the quota is met; with a further follow up of up to 12 weeks post-surgical intervention.

Patients meeting the inclusion criteria will be informed of the study and once agreement to participate is obtained, will be invited to a private room to go through the consenting process. All consents will be done by the Research Assistant at that clinical visit. The time taken to perform the surgery after consent will be based on surgical time availability and patient finances, both of which should not distort standard of care or patient outcomes. All data obtained will be digitized and stored on a secure encrypted hard drive stored in the office of the Principal Investigator only accessible by the research team.

Procedure Administration The procedure will take place in the Main Operating Theatre. Patients will be randomized by the online randomization tool and assigned a study ID number, and a study group. This will be logged by the Research Assistant and information kept stored in the principal investigator's office computer. The participant will be transported to the operating theatre with a sealed envelope affixed to their docket containing that study ID number issued.

The Research Assistant will collect the envelop and reference the number with a randomization chart provided syncing the groups assigned.

The Research Assistant in a separate designated room will aspirate either TXA (10 mL, 1g) or saline (10 mL) alone dependent on the number given by the randomization tool. The aspirate will be placed in a marked syringe and given to the patient via intravenous transfusion of 100 mLs saline over a 10-minute period.

All patients to undergo Arthroscopic ACL reconstruction after being assigned to their respective groups and randomized intervention, will receive TXA (10 mL, 1g) in 100 mLs of saline. The control group will receive 110 mLs of saline total 10mins prior to surgery at the same rate and the same route. This will be administered by the anesthetic team under the guidance of the independent team Research Assistant. The surgeon and patient will be blinded, however the anesthesiologist will not be blinded.

Surgical Technique All patients will be positioned supine and administered spinal anesthesia. In all cases the application of a pneumatic torniquet will be applied to the proximal thigh after induction of anesthesia but will not be inflated for the group receiving TXA. Dependent on the randomized groups assigned; The standard torniquet pressure of 300 mm Hg will only be inflated for persons assigned to the torniquet group who will receive normal saline intravenously. Only the Research Assistant and the anesthetic staff will be aware of whether inflation of torniquet was applied. No other methods of hemostasis will be used for example, e.g., intra-articular cautery, Saline diluted epinephrine aliquots or 4 °C normal saline irrigation.

Postoperative Care Post ACL harvesting, the patients will undergo the standard two portal knee arthroscopy with a pressure pump injector set at the standard 30 psi. Visibility will be assessed using a 3 pronged questionnaire about intraoperative visibility by the main surgeon (7) which was shown to be better validated and with less inter-observer bias than 10-point scoring systems, with 3 being complete lack of vision and 1 being complete clarity (Appendix E).

The proposed start time of the study is July 2024.

Assessment of Risks and Benefits This research is a moderate risk study. The potential risks of tranexamic and physiological risk of thromboembolic phenomenon although proven highly unlikely must be considered (38).

Pneumatic torniquet being used as a standard of care in ACL reconstruction does have its negative such as compartment syndrome, neurapraxia due to prolonged compression, quadriceps lag and prolonging rehabilitation (39). The study has strict guidelines to ensure safety, hence the recommended 300 mm Hg pressure for inflation.

The benefit of this study is to gain the awareness of tranexamic acids use its vast potential as an alternate alternative standard of care in improving visibility during arthroscopic ACL reconstructive surgery.

No patient will be coerced to participate. No intervention deemed clinically necessary would be withheld from any participant or any who refuse consent.

Confidentiality Each patient will be assigned a study number which will be logged and kept by the research team. Information will be stored on a storage device that will be password protected stored in the principal investigator's office and accessed only by the research team.

Compensation and payments There will be no waiver of clinic fees as outpatient department clinic reviews at 2 weeks and 3 months are the normal standard of care for all patients. No compensation will be given to patients who consent to participate in the study.

Funding Funding if needed for this project will be provided by the research team. (Appendix C)

Expected Outcome Findings of the study will be used for publications and/or presentations both locally and internationally.

Ethical Considerations Ethical guidelines will be adhered to following the approval of the Mona Campus Research Ethics Committee (MCREC). Patients will be given a chance to ask questions and consider their participation freely during the informed consent process. Patients will be advised of their right to withdraw from the study at any point without the need for an explanation and care will not be withheld from those who do not participate. Patients' autonomy and dignity will be always protected.

Conflict of Interest There is no conflict of interest with the manufacturers of the drug being studied

Fair Selection of Subjects Subjects will be selected only because of the specific problem under investigation (i.e. patients with the condition Complete ACL rupture), being seen in the Orthopedic Outpatient Department at the UHWI or privately.) No participant in this study will be chosen due to easy availability, diminished autonomy, or social bias.

Limitations:

The foreseeable limitation to the study is the surgeon not being blinded can be prevented by:

1. Allowing main surgeons in the Operating theatre after all interventions and controls have been performed.
2. Post preparation of the surgical field with sterile drapes. However, if these measures fail to prevent blinding mitigating measures include

1. Patient data would have to discarded. 2. A second surgeon as experienced absent during intervention or control would assess visual clarity as well based on the scale provided.

Impact of the study:

The results will be disseminated at academic meetings, international presentations and published in a peer review journal.

ELIGIBILITY:
Inclusion Criteria:

* All patients with complete ACL tears requiring reconstruction for the first time.
* Ages >18

Exclusion Criteria:

* Dementia or any patient with cognitive impairment.
* Patients with previous functional disabilities (Patients with functional disabilities affecting the lower limb such as stroke, neuromuscular disorders or any pathology limiting Knee range of motion can cause abnormalities within the joint enabling scaring, fibrosis or even hypoplastic degenerating tissue. These features may alter the vascularity and directly affect visual clarity)
* Bleed disorders or coagulopathies.
* Sickle Cell Disease, liver, or renal failure.
* Multi- ligamentous knee injuries.
* Anticoagulant therapy.
* Revision ACL reconstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Grading TXA | The questionnaire will be administered to the surgeon right after surgery is completed.
  The grading allotted to patients treated with tranexamic acid assed by the Arthroscopic visual clarity scale.
Grading Tourniquet | The questionnaire will be administered to the surgeon right after surgery is completed.
  The Grading given to patients treated with Pneumatic torniquet assessed by the Arthroscopic Visual clarity scale
Grading Tourniquet vs TXA | The questionnaire will be administered to the surgeon right after surgery is completed.
  The grading given to patients treated with TXA vs Pneumatic torniquet assessed by the arthroscopic visual clarity scale

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of the West Indies, Department of Surgery, Kingston, Jamaica, Jamaica

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choudhary A, Kanodia N, Agrawal S, Bhasin VB, Singh A. Tourniquet Use in Arthroscopic ACL Reconstruction: A Blinded Randomized Trial. Indian J Orthop. 2020 Sep 12;55(2):384-391. doi: 10.1007/s43465-020-00250-z. eCollection 2021 Apr. PMID 33927817
- [Background] Ockerman A, Vanassche T, Garip M, Vandenbriele C, Engelen MM, Martens J, Politis C, Jacobs R, Verhamme P. Tranexamic acid for the prevention and treatment of bleeding in surgery, trauma and bleeding disorders: a narrative review. Thromb J. 2021 Aug 11;19(1):54. doi: 10.1186/s12959-021-00303-9. PMID 34380507
- [Background] Hoogeslag RA, Brouwer RW, van Raay JJ. The value of tourniquet use for visibility during arthroscopy of the knee: a double-blind, randomized controlled trial. Arthroscopy. 2010 Sep;26(9 Suppl):S67-72. doi: 10.1016/j.arthro.2009.12.008. Epub 2010 May 13. PMID 20810094
- [Background] Smith TO, Hing CB. A meta-analysis of tourniquet assisted arthroscopic knee surgery. Knee. 2009 Oct;16(5):317-21. doi: 10.1016/j.knee.2009.01.004. Epub 2009 Feb 23. PMID 19239987
- [Background] Stefan AM, Gronau QF, Schonbrodt FD, Wagenmakers EJ. A tutorial on Bayes Factor Design Analysis using an informed prior. Behav Res Methods. 2019 Jun;51(3):1042-1058. doi: 10.3758/s13428-018-01189-8. PMID 30719688
- [Background] Robert C, Chopin N, Rousseau J, Bernardo J, Gelman A, Kass R, et al. Harold Jeffreys's Theory of Probability Revisited. 2008.
- [Background] Vargha A, Delaney H. A Critique and Improvement of the "CL" Common Language Effect Size Statistics of McGraw and Wong. Journal of Educational and Behavioral Statistics - J EDUC BEHAV STAT. 2000;25.
- [Background] Aziz Catalttepe KO. The effect of a single dose of intravenous tranexamic acid on visual clarity in knee arthroscopic meniscectomy without a tourniquet
- [Background] Patel NK, Johns W, Vedi V, Langstaff RJ, Golladay GJ. Tourniquet and tranexamic acid use in total knee arthroplasty. Arthroplast Today. 2020 Apr 28;6(2):246-250. doi: 10.1016/j.artd.2020.02.007. eCollection 2020 Jun. PMID 32577472
- [Background] Jennings JD, Solarz MK, Haydel C. Application of Tranexamic Acid in Trauma and Orthopedic Surgery. Orthop Clin North Am. 2016 Jan;47(1):137-43. doi: 10.1016/j.ocl.2015.08.014. PMID 26614928
- [Background] Hofmann A, Ozawa S, Farrugia A, Farmer SL, Shander A. Economic considerations on transfusion medicine and patient blood management. Best Pract Res Clin Anaesthesiol. 2013 Mar;27(1):59-68. doi: 10.1016/j.bpa.2013.02.001. PMID 23590916
- [Background] Marik PE, Corwin HL. Efficacy of red blood cell transfusion in the critically ill: a systematic review of the literature. Crit Care Med. 2008 Sep;36(9):2667-74. doi: 10.1097/CCM.0b013e3181844677. PMID 18679112
- [Background] Zollo RA, Eaton MP, Karcz M, Pasternak R, Glance LG. Blood transfusion in the perioperative period. Best Pract Res Clin Anaesthesiol. 2012 Dec;26(4):475-84. doi: 10.1016/j.bpa.2012.10.001. PMID 23351234
- [Background] Han C, Liu M, Lian X, Sun T, Yan S, Bai X, Gan D, Leng B, Qiu Y, Ren Y. Tranexamic acid use in arthroscopic rotator cuff repair is an effective and safe adjunct to improve visualization: a systematic review and meta-analysis. J Shoulder Elbow Surg. 2023 Nov;32(11):2389-2399. doi: 10.1016/j.jse.2023.06.013. Epub 2023 Jul 17. PMID 37468032
- [Background] Kawaguchi S, Fukuta S, Kano M, Sairyo K. Reduction of perioperative blood loss and operating time for arthroscopic rotator cuff repair by intravenous administration of tranexamic acid. Asia Pac J Sports Med Arthrosc Rehabil Technol. 2023 Feb 7;31:6-10. doi: 10.1016/j.asmart.2023.01.001. eCollection 2023 Jan. PMID 36820053
- [Background] Ersin M, Demirel M, Buget MI, Edipoglu IS, Atalar AC, Ersen A. The effect of intravenous tranexamic acid on visual clarity during arthroscopic rotator cuff repair: A randomized, double-blinded, placebo-controlled pilot study. Acta Orthop Traumatol Turc. 2020 Nov;54(6):572-576. doi: 10.5152/j.aott.2020.19164. PMID 33423986
- [Background] Liu YF, Hong CK, Hsu KL, Kuan FC, Chen Y, Yeh ML, Su WR. Intravenous Administration of Tranexamic Acid Significantly Improved Clarity of the Visual Field in Arthroscopic Shoulder Surgery. A Prospective, Double-Blind, and Randomized Controlled Trial. Arthroscopy. 2020 Mar;36(3):640-647. doi: 10.1016/j.arthro.2019.10.020. Epub 2019 Dec 20. PMID 31870749
- [Background] Dugani S, Wasan KM, Kissoon N. World Health Organization and Essential Medicines. J Pharm Sci. 2018 May;107(5):1261-1262. doi: 10.1016/j.xphs.2017.12.019. Epub 2017 Dec 24. PMID 29277641
- [Background] Haratian A, Shelby T, Hasan LK, Bolia IK, Weber AE, Petrigliano FA. Utilization of Tranexamic Acid in Surgical Orthopaedic Practice: Indications and Current Considerations. Orthop Res Rev. 2021 Oct 19;13:187-199. doi: 10.2147/ORR.S321881. eCollection 2021. PMID 34703327
- [Background] Pabinger I, Fries D, Schochl H, Streif W, Toller W. Tranexamic acid for treatment and prophylaxis of bleeding and hyperfibrinolysis. Wien Klin Wochenschr. 2017 May;129(9-10):303-316. doi: 10.1007/s00508-017-1194-y. Epub 2017 Apr 21. PMID 28432428
- [Background] Hao S, Li H, Liu S, Meng S, Zhang X, Wang L, Yang H, Zhang L, Dong S. The effect of intravenous unit-dose tranexamic acid on visible and hidden blood loss in posterior lumbar interbody fusion: a randomized clinical trial. Sci Rep. 2023 Mar 22;13(1):4714. doi: 10.1038/s41598-022-27307-3. PMID 36949108
- [Background] Vrontis K, Tsinaslanidis G, Drosos GI, Tzatzairis T. Perioperative Blood Management Strategies for Patients Undergoing Total Hip Arthroplasty: Where Do We Currently Stand on This Matter? Arch Bone Jt Surg. 2020 Nov;8(6):646-655. doi: 10.22038/abjs.2020.45651.2249. PMID 33313343
- [Background] Picetti R, Shakur-Still H, Medcalf RL, Standing JF, Roberts I. What concentration of tranexamic acid is needed to inhibit fibrinolysis? A systematic review of pharmacodynamics studies. Blood Coagul Fibrinolysis. 2019 Jan;30(1):1-10. doi: 10.1097/MBC.0000000000000789. PMID 30585835
- [Background] Yaghmour KM, Al-Khateeb H. Anterior cruciate ligament reconstruction without the use of a tourniquet. Ann R Coll Surg Engl. 2019 Feb;101(2):123-125. doi: 10.1308/rcsann.2018.0197. Epub 2018 Nov 1. PMID 30381954
- [Background] Carter KB, Shaw A, Telfer AB. Tourniquets for surgery: safety aspects. J Med Eng Technol. 1983 May-Jun;7(3):136-9. doi: 10.3109/03091908309032577. PMID 6876134
- [Background] Liu D, Graham D, Gillies K, Gillies RM. Effects of tourniquet use on quadriceps function and pain in total knee arthroplasty. Knee Surg Relat Res. 2014 Dec;26(4):207-13. doi: 10.5792/ksrr.2014.26.4.207. Epub 2014 Dec 2. PMID 25505702
- [Background] Masri BA, Eisen A, Duncan CP, McEwen JA. Tourniquet-induced nerve compression injuries are caused by high pressure levels and gradients - a review of the evidence to guide safe surgical, pre-hospital and blood flow restriction usage. BMC Biomed Eng. 2020 May 28;2:7. doi: 10.1186/s42490-020-00041-5. eCollection 2020. PMID 32903342
- [Background] Atisuksma ID, Rhatomy S, Dewo P. A tourniquet-less technique using saline epinephrine irrigation system in an arthroscopic ACL reconstruction in patient with history of popliteal artery ligation. Int J Surg Case Rep. 2018;53:157-162. doi: 10.1016/j.ijscr.2018.10.040. Epub 2018 Nov 1. PMID 30396128
- [Background] Derriks JHG, Hilgersom NFJ, Middelkoop E, Samuelsson K, van den Bekerom MPJ. Electrocautery in arthroscopic surgery: intra-articular fluid temperatures above 43 degrees C cause potential tissue damage. Knee Surg Sports Traumatol Arthrosc. 2020 Jul;28(7):2270-2278. doi: 10.1007/s00167-019-05574-4. Epub 2019 Jun 27. PMID 31250052
- [Background] Olszewski AD, Jones R, Farrell R, Kaylor K. The effects of dilute epinephrine saline irrigation on the need for tourniquet use in routine arthroscopic knee surgery. Am J Sports Med. 1999 May-Jun;27(3):354-6. doi: 10.1177/03635465990270031501. PMID 10352773
- [Background] Hsiao MS, Kusnezov N, Sieg RN, Owens BD, Herzog JP. Use of an Irrigation Pump System in Arthroscopic Procedures. Orthopedics. 2016 May 1;39(3):e474-8. doi: 10.3928/01477447-20160427-01. Epub 2016 May 2. PMID 27135450
- [Background] Li S, A L. The hidden blood loss and its factors in patients undergoing minimally invasive knee arthroscopy. Front Surg. 2022 Aug 30;9:944481. doi: 10.3389/fsurg.2022.944481. eCollection 2022. PMID 36111226
- [Background] Palmer W, Critchlow A, Mansingh A. Return to Sports and Functional Outcome after Primary Anterior Cruciate Ligament Reconstruction in Jamaica. Sports Nutrition and Therapy. 2016;1.
- [Background] van Montfoort DO, van Kampen PM, Huijsmans PE. Epinephrine Diluted Saline-Irrigation Fluid in Arthroscopic Shoulder Surgery: A Significant Improvement of Clarity of Visual Field and Shortening of Total Operation Time. A Randomized Controlled Trial. Arthroscopy. 2016 Mar;32(3):436-44. doi: 10.1016/j.arthro.2015.08.027. PMID 26524933
- [Background] Biz C, Cigolotti A, Zonta F, Belluzzi E, Ruggieri P. ACL reconstruction using a bone patellar tendon bone (BPTB) allograft or a hamstring tendon autograft (GST): a single-center comparative study. Acta Biomed. 2019 Dec 5;90(12-S):109-117. doi: 10.23750/abm.v90i12-S.8973. PMID 31821294
- [Background] Domnick C, Raschke MJ, Herbort M. Biomechanics of the anterior cruciate ligament: Physiology, rupture and reconstruction techniques. World J Orthop. 2016 Feb 18;7(2):82-93. doi: 10.5312/wjo.v7.i2.82. eCollection 2016 Feb 18. PMID 26925379
- [Background] Gans I, Retzky JS, Jones LC, Tanaka MJ. Epidemiology of Recurrent Anterior Cruciate Ligament Injuries in National Collegiate Athletic Association Sports: The Injury Surveillance Program, 2004-2014. Orthop J Sports Med. 2018 Jun 13;6(6):2325967118777823. doi: 10.1177/2325967118777823. eCollection 2018 Jun. PMID 29977938
- [Background] Wojtys EM, Brower AM. Anterior cruciate ligament injuries in the prepubescent and adolescent athlete: clinical and research considerations. J Athl Train. 2010 Sep-Oct;45(5):509-12. doi: 10.4085/1062-6050-45.5.509. No abstract available. PMID 20831399